CLINICAL TRIAL: NCT04888481
Title: 68Ga-HA-DOTATATE Imaging of Suspected Somatostatin Receptor Positive Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CC-19-0369
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — 68Ga-DOTA-iodo-Tyr(3)-octreotate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-HA-DOTATATE PET/CT scan (Experimental): 2.64 MBq/kg (minimum 37 MBq, maximum 250 MBq) 68Ga-HA-DOTATATE intravenous single-dose administration for PET/CT imaging
  Interventions: Drug: 68Ga-HA-DOTATATE

INTERVENTIONS:
Drug: 68Ga-HA-DOTATATE — Tracer injection

SUMMARY:
Somatostatin receptor (SSR) imaging is a critical component of clinical care for many patients being investigated for or with confirmed SSR positive tumors. In the past, 111In-octreotide imaging has been used for this purpose but it has been recently supplanted globally by SSR positron emission tomography (PET) imaging due to better image quality and higher diagnostic accuracy.

This study will assess the safety and diagnostic effectiveness of 68Ga-HA-DOTATATE produced a the Edmonton Radiopharmaceutical Centre (ERC).

DETAILED DESCRIPTION:
A single centre non-randomized, non-blinded phase II prospective cohort study evaluating the safety and efficacy of 68Ga-HA-DOTATATE PET/CT imaging in patients with known or suspected somatostatin receptor positive tumors.

Up to 600 scans will be included over 6 years. All patient ages (pediatric and adult) will be included. Individual patients may have more than one scan during the study period.

Safety evaluation will consist of an adverse event assessment whil in the Nuclear Medicine department at the University of Alberta Hospital. Efficacy evaluation will consist of a comparison to CT and/or MRI accuracy based on 1 year follow-up clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known or clinically suspected somatostatin receptor positive tumors including but not limited to: gastrointestinal neuroendocrine tumors, pancreatic neuroendocrine tumors, pulmonary neuroendocrine tumors, neuroendocrine tumors - primary unknown, pheochromocytoma, paraganglioma, medullary thyroid cancer, medulloblastoma, meningioma
* A standard clinical CT or MRI is obtained within 6 months of enrollment
* Ability to provide written informed consent prior to participation in the study (participant or if required a legal medical decision maker)

Exclusion Criteria:

* Weight > 225 kg (weight limit of the PET/CT scanner)
* Inability to scan (ie. extreme claustrophobia) or inability to lie still for imaging
* Any additional medical condition, serious inter-current illness, or other extenuating circumstance that, in the opinion of the investigator or attending department physician, may significantly interfere with study performance or interpretation
* Previous allergic reaction to DOTATATE or somatostatin analogues
* Lack of intravenous access

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy - sensitivity | 1 year post-scan
  Sensitivity of 68Ga-HA-DOTATATE PET/CT compared to 1 year clinical follow-up
Efficacy - specificity | 1 year post-scan
  Specificity of 68Ga-HA-DOTATATE PET/CT compared to 1 year clinical follow-up

SECONDARY OUTCOMES:
Safety - adverse events - immediate | Immediately (within 15 minutes) after tracer injection
  Assessment of adverse events immediately after tracer injection
Safety - adverse events - post-scan | Immediately (within 15 minutes) after PET/CT scan; 60 to 100 minutes after tracer injection
  Assessment of adverse events immediately after PET/CT scan
Safety - adverse events - delayed | 10 days after tracer injection
  Self-reporting of possible adverse events after leaving the PET department

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Abele, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No